CLINICAL TRIAL: NCT04624256
Title: Germline DNA-Based Radiosensitivity Biomarker Influence on Toxicity Following Prostate Radiotherapy
Brief Title: Germline DNA-Based Radiosensitivity Biomarker Influence on Toxicity Following Prostate Radiotherapy, GARUDA Trial
Acronym: GARUDA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: MiraDX (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-001386; NCI-2020-07928 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-10-26; First posted 2020-11-10 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Prostate Adenocarcinoma; Stage I Prostate Cancer American Joint Committee on Cancer (AJCC) v8; Stage II Prostate Cancer AJCC v8; Stage IIA Prostate Cancer AJCC v8; Stage IIB Prostate Cancer AJCC v8; Stage IIC Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiation Dose Hypofractionation; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (radiotherapy, genomic DNA testing) (Experimental): Patients undergo SBRT per standard of care, then undergo collection of cheek swab and blood samples for the analysis of germline biomarkers. Afterwards, patients and their physicians engage in discussion about which form of radiotherapy to proceed with. Based on the decision, patients predicted to be at low risk of toxicity with SBRT continue to receive SBRT over 14 days while patients predicted to be at high risk of toxicity with SBRT will be counseled to undergo either conventionally fractionated radiotherapy over 63-70 days, moderate hypofractionated radiotherapy over 28-35 days, or may opt to still receive SBRT over 14 days per standard of care.
  Interventions: Procedure: Discussion; Radiation: Hypofractionated Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Procedure: Discussion — Patients and physicians engage in discussion
  Other Names: Discuss
Radiation: Hypofractionated Radiation Therapy — Undergo conventional hypofractionated radiation therapy
  Other Names: Hypofractionated Radiotherapy; hypofractionation
Radiation: Hypofractionated Radiation Therapy — Undergo moderate hypofractionated radiation therapy
  Other Names: Hypofractionated Radiotherapy; hypofractionation
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This trial studies the changes in long-term physician-scored genitourinary toxicity achieved in prostate cancer patients eligible for stereotactic radiation therapy when both patients and physicians have access to convincing but non-validated germline signature that can characterize patients as having a low or high risk of developing toxicity after radiation therapy. The information learned from this study may guide patients' and physicians' decisions on radiotherapy fractionation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the impact on the 5-year cumulative incidence of late grade >= 2 genitourinary (GU) physician-scored toxicity, as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 scale, caused by presenting both the physicians and patients with the results of a non-prospectively validated biomarker panel that dichotomizes any given patient into having a high versus a low risk of late grade >= 2 GU physician-scored toxicity following stereotactic body radiotherapy (SBRT).

SECONDARY OBJECTIVES:

I. To determine the late grade >= 2 genitourinary (GU) physician-scored toxicity, as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 scale, in patients who test positive for the biomarker.

II. To determine the late grade >= 2 genitourinary (GU) physician-scored toxicity, as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 scale, in patients who test negative for the biomarker.

III. To observe the proportions of patients who choose to receive conventionally fractionated radiotherapy, moderately hypofractionated radiotherapy, and SBRT, based on being positive or negative for the biomarker thought to predict for late grade >= 2 GU toxicity.

IV. To determine the 5-year cumulative incidence of late grade >= 2 gastrointestinal (GI) physician-reported toxicity, as assessed by the CTCAE version 4.03 scale, following the same intervention as for the primary objective.

V. To determine the incidence of acute grade >= 2 GU and GI toxicity as assessed by the CTCAE version 4.03 scale, following the same intervention as for the primary objective.

VI. To quantify the temporal changes in patient-reported quality of life (QOL) outcomes, as assessed by the Expanded Prostate Cancer Index-26 (EPIC-26), International Prostate Symptom Scores (IPSS), and Sexual Health Inventory for Men (SHIM) QOL indices, following the same intervention as for the primary objective.

OUTLINE:

Patients planning to undergo SBRT per standard of care undergo collection of cheek swab and blood samples for the analysis of germline biomarkers. Afterwards, patients and their physicians engage in discussion about which form of radiotherapy to proceed with. Based on the decision, patients predicted to be at low risk of toxicity with SBRT continue to receive SBRT over 14 days while patients predicted to be at high risk of toxicity with SBRT will be counseled to undergo either conventionally fractionated radiotherapy over 63-70 days, moderate hypofractionated radiotherapy over 28-35 days, or may opt to still receive SBRT over 14 days per standard of care.

After completion of radiotherapy treatment, patients are followed up at 1 ,3, 6, 9, 12, 18, and 24 months, and then every 6 months for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, clinical localized adenocarcinoma of the prostate
* No evidence of disease beyond the prostate and/or seminal vesicles (i.e., no suspicious pelvic lymph nodes or presence of metastatic disease outside the pelvis)
* Staging workup as recommended by the National Comprehensive Cancer Network (NCCN) on the basis of risk grouping:

  * Low risk: No staging workup required
  * Favorable intermediate-risk: computed tomography (CT) abdomen/pelvis only if Memorial Sloan Kettering Cancer Center (MSKCC) nomogram predicts > 10% probability of lymph node involvement (note: CT simulation scan will count as a CT abdomen/pelvis)
  * Unfavorable intermediate-risk: technetium bone scan, CT abdomen/pelvis if MSKCC nomogram predicts > 10% probability of lymph node involvement (note: CT simulation scan will count as a CT abdomen/pelvis)
  * High-risk: technetium bone scan, CT abdomen/pelvis if MSKCC nomogram predicts > 10% probability of lymph node involvement (note: CT simulation scan will count as a CT abdomen/pelvis) =
  * Advanced imaging studies (i.e. prostate specific membrane antigen [PSMA] positron emission tomography [PET] and Axumin scan) can supplant a bone scan if performed first
* Ability to understand, and willingness to sign, the written informed consent

Exclusion Criteria:

* Patients with neuroendocrine or small cell carcinoma of the prostate
* Patients with any evidence of distant metastases. Note, evidence of lymphadenopathy below the level of the renal arteries can be deemed loco regional per the discretion of the investigator
* Prior whole-gland cryosurgery, high-intensity focused ultrasound (HIFU) or brachytherapy of the prostate
* Prior pelvic radiotherapy
* History of Crohn's disease, ulcerative colitis, or ataxia telangiectasia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
5-year cumulative incidence of late grade >= 2 physician-scored genitourinary toxicity | Up to 5 years
  Assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 scale, stratified by positive or negative status for the biomarker thought to predict for late grade >= 2 genitourinary (GU) toxicity.

SECONDARY OUTCOMES:
5-year biochemical recurrence-free survival | Up to 5 years
  Will be estimated by the Kaplan-Meier method, with biochemical recurrence (BCR) defined as serum prostate specific antigen (PSA) levels that are 2 ng/mL higher than the nadir PSA achieved after magnetic resonance imaging-guided stereotactic body radiation therapy (SBRT).
Rate of acute grade >= 2 genitourinary and gastrointestinal physician-scored toxicity | Up to the first 90 days after radiotherapy
  Assessed by the CTCAE version 4.03 scale, based on being positive or negative for the biomarker thought to predict for late grade >= 2 GU toxicity. The timeframe will be restricted to the first 90 days after radiotherapy.
Rate of acute grade >= 2 gastrointestinal physician-scored toxicity | Up to the first 90 days after radiotherapy (acute).
  Assessed by the CTCAE version 4.03 scale, based on being positive or negative for the biomarker thought to predict for late grade >= 2 GU toxicity.
5-year cumulative incidence of Late grade >= 2 GU physician-scored toxicity | Up to 5 years
  Assessed by the CTCAE version 4.03 scale, in patients who test positive or negative for the biomarker.
Proportions of patients who choose to receive radiation treatment | Up to 5 years
  Will analyze the proportions of patients who choose to receive conventionally fractionated radiotherapy, moderately hypofractionated radiotherapy, and SBRT, based on being positive or negative for the biomarker thought to predict for late grade >= 2 GU toxicity.
Change in patient-reported urinary quality of life | Baseline up to 5 years
  Will be obtained depending on the instrument used. For the Expanded Prostate Cancer Index-26 instrument, these will be represented by changes from baseline in the urinary symptom domain. The scores will range from 0-100, with a higher number indicating a better quality of life. Changes will be analyzed with respect to whether they represent minimally important differences, based on approved thresholds in the literature.
Change in patient-reported bowel quality of life | Baseline up to 5 years
  Will be obtained depending on the instrument used. For the Expanded Prostate Cancer Index-26 instrument, these will be represented by changes from baseline in the bowel domain. The scores will range from 0-100, with a higher number indicating a better quality of life. Changes will be analyzed with respect to whether they represent minimally important differences.
Change in patient-reported sexual quality of life outcome | Baseline up to 5 years
  will be assessed by the International Prostate Symptom Scores (I-PSS) instrument by five years. Scoring is from 1 - 35, a higher number is worse outcome.
Change in patient-reported sexual quality of life by the Sexual Health Inventory for Men instrument by five years | Baseline up to 5 years
  Will be represented by changes from baseline in the urinary incontinence and urinary obstruction domains on the Sexual Health Inventory for Men instrument (SHIM). coring from 1-25, higher number is better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Amar Kishan, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States